CLINICAL TRIAL: NCT06514339
Title: Evidence-based Evaluation and Mechanism of Shenhuang Granules in the Treatment of Sepsis: a Randomized, Double-blind, Placebo-controlled, Effective Clinical Trial
Brief Title: Evidence-based Evaluation and Mechanism of Shenhuang Granules in the Treatment of Sepsis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang University (Other); Red Cross Hospital, Hangzhou, China (Other); Ningbo Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-KLS-234-02
Record Dates: First submitted 2024-06-19; First posted 2024-07-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
Keywords: Sepsis; Shenhuang granules; Evidence-based evaluation; Effect mechanism research
MeSH Terms: conditions — Sepsis | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Intervention Model Description: The researchers were randomly assigned to either a trial or a control group. Experimental group: sepsis cluster therapy + Shenhuang granules, course of 5 days. For the treatment of sepsis cluster, refer to the 2021 International Guidelines for Severe Sepsis and Septic Shock. Shenhuang Granules (Tianjin Hongri Pharmaceutical Co., LTD.) : 2 times a day, 1 pack each time, 100ml of warm water (temperature about 40°C) after dissolution, oral or nasal feeding (stomach tube or intestinal tube).
  Control group: sepsis cluster therapy + placebo for 5 days. For the treatment of sepsis cluster, refer to the 2021 International Guidelines for Severe Sepsis and Septic Shock. Placebo (Tianjin Hongri Pharmaceutical Co., LTD.) : After dissolution of 100ml warm water (temperature about 40°C) in 1 pack twice a day, oral or nasal feeding (gastric tube or intestinal tube).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will adopt the block randomization method to randomly assign qualified subjects to the test group or the control group in a ratio of 1:1. A central randomization system was used for randomization and drug distribution management. From randomization until the database is locked, subjects, investigators, data analysts, sponsors, and all medical personnel involved in the treatment or clinical evaluation will remain blind to the reality of the treatment.
  The random number table (blind bottom) used in this study will be generated by the randomization specialist and imported into the system. The random number is reproducible. The relationship between the experimental group drug or the control group simulated drug and the subjects was represented by random number and drug number. The blind bottom is kept by the randomisation Specialist and remains unknown to both subjects and investigators throughout the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Sepsis cluster therapy + Shenhuang granules for 5 days. For the treatment of sepsis cluster, refer to the 2021 International Guidelines for Severe Sepsis and Septic Shock. Shenhuang Granules (Tianjin Hongri Pharmaceutical Co., LTD.) : 2 times a day, 1 pack each time, 100ml of warm water (temperature about 40°C) after dissolution, oral or nasal feeding (stomach tube or intestinal tube).
  Interventions: Drug: shenhuang granule
- Control group (Sham Comparator): Sepsis cluster therapy + placebo for 5 days. For the treatment of sepsis cluster, refer to the 2021 International Guidelines for Severe Sepsis and Septic Shock. Placebo (Tianjin Hongri Pharmaceutical Co., LTD.) : After dissolution of 100ml warm water (temperature about 40°C) in 1 pack twice a day, oral or nasal feeding (gastric tube or intestinal tube).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: shenhuang granule — Traditional Chinese medicine compound "Shenhuang Granules" is developed by Professor Fang Bangjiang, a scholar in the team of Qi-Huang, which is composed of ginseng, rhubarb, dandelion, etc., with the effect of Fuzheng Guben, clearing heat and detoxification, promoting qi and promoting blood and detumification.
  Other Names: Tianjin Hongri Pharmaceutical Co., LTD
  Arms: Treatment group
Drug: placebo — Placebo was provided by Tianjin Hongri Pharmaceutical Co., LTD., and was given orally or nasally (through gastric tube or intestinal tube) after dissolution of 100ml warm water (temperature about 40°) in 1 package twice a day.
  Other Names: Tianjin Hongri Pharmaceutical Co., LTD
  Arms: Control group

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by the body's dysfunctional response to infection, most patients require treatment in the ICU, and is the leading cause of death worldwide. Over the years, the development of new drugs for the treatment of sepsis has failed without significant benefit in reducing mortality, and there is currently no effective drug treatment. Therefore, sepsis is a serious disease threatening the life and health of patients, causing a huge burden to society, and is a major problem in the medical field.

The pathogenesis of sepsis is complicated, and immune imbalance is the key mechanism. Suppression of host immune function may be the root cause of the increase in the long-term mortality of sepsis. Bidirectional immune regulation may be an important treatment plan to improve the survival rate and quality of life of sepsis patients. In recent years, the contribution of traditional Chinese medicine to sepsis has been highly valued at home and abroad. The treatment of sepsis by traditional Chinese medicine mainly plays the role of bidirectional immune regulation by dispelling the evil and supporting the right. Our team has achieved some results in the diagnosis and treatment of sepsis by using traditional Chinese medicine. Supported by National Natural Science Foundation of China (81774070). The team also found that magnolol can inhibit intestinal mucosal inflammation in sepsis, which was also supported by the National Natural Science Foundation of China (82174178). The team of Qhuang scholars inherit the academic experience of Zhu Liangchun, the master of Chinese medicine, warm and hot disease need not be limited to the law of wei, qi, ying, blood transmission, that is, the disease can be solved both outside and inside, breaking the three bans of warm and cold disease. On the basis of inheriting Zhu Liangchun's academic theory, the author put forward the early treatment rule of "truncation and reversal", and used to cleanse the "poison" and "save Yin" in the early stage of sepsis to quickly truncate the malignant development trend of sepsis. In the COVID-19 epidemic, we have found that patients with COVID-19 sepsis have "acute deficiency syndrome" in the early stage of clinical syndrome, which is an important factor leading to death. The clinical efficacy and mechanism of "Shenhuang Granules" in sepsis caused by non-novel coronavirus infection such as bacteria need to be further studied.

DETAILED DESCRIPTION:
1. Baseline data: patient's name, gender, age, enrollment diagnosis, sepsis diagnosis time, combined underlying disease, allergy history, personal history, body temperature, respiration, heart rate, blood pressure, blood oxygen saturation and other vital signs.
2. Primary outcome measure: 28-day mortality
3. Secondary outcome indicators:

   A. Total length of stay and ICU stay B. Total hospitalization costs and ICU hospitalization costs C. Overall mortality and ICU mortality D.28 days cumulative no mechanical ventilation time E. Information of TCM syndrome such as tongue and pulse on day 0 and day 5-7 F. TCM symptom scores on days 0 and 5-7 G. SOFA score and APACHE II score on days 0 and 5-7.
4. Other observation indicators (day 0 and 7) :

   A. Inflammatory markers: WBC, percentage of neutrophils, CRP, PCT, tumor necrosis factor (TNF-α), interleukin-6 (IL-6), interleukin-10 (IL-10); B. Main organ function indicators: BNP, TnI, creatinine, urea nitrogen, total bilirubin, direct bilirubin, indirect bilirubin, AST, ALT, arterial lactic acid; C. Coagulation indicators: PT, APTT; D. Immune function: absolute number of lymphocytes, number of CD4+T cells, number of CD8+T cells, number of B cells, number of NK cells.
5. Safety indicators: adverse reaction symptoms or adverse events (such as allergies).

   If you need to collect stool and blood samples, you also need to observe the following indicators, if not, please ignore.
6. Metabolomic study: Serum samples from day 0 and day 5-7 were collected for the study of the main functional components of Shenhuang granules and metabolomic analysis;
7. Intestinal microecology study: Stool samples from day 0 and day 5-7 were collected for intestinal microecology study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Meet the diagnostic criteria of sepsis 3.0 guidelines
* Sign informed consent.

Exclusion Criteria:

* Liver or kidney single SOFA score ≥3 points of liver and kidney dysfunction
* Death is expected within 48 hours, or SOFA≥15 points, or APACHE II ≥30 points, or the patient refuses active treatment
* Patients with allergic reactions to traditional Chinese medicine
* Patients treated with chemotherapy or radiotherapy or high-dose immunosuppressants within the last 1 month
* Participants in other clinical trials at the same time or within 30 days
* Pregnant and lactating women
* Patients with severe gastrointestinal bleeding, intestinal obstruction, or severe intraperitoneal pressure elevation (IAP≥20mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality rate | 28-day
  The proportion of deaths due to illness within 28 days after treatment began

SECONDARY OUTCOMES:
Total length of stay and ICU stay | 7 day after treatment，14 day after treatment，28 day after treatment
  Total length of stay and length of stay in ICU
Total hospitalization costs and ICU hospitalization costs | 7 day after treatment，14 day after treatment，28 day after treatment
  The patient's total hospitalization costs and hospitalization costs in the ICU
Overall mortality and ICU mortality | 7 day after treatment，14 day after treatment，28 day after treatment
  The proportion of patients who died during their total hospital stay and the proportion of patients who died during their ICU stay were included
28 days cumulative no mechanical ventilation time | 28 day after treatment
  The total time the patient spent without mechanical ventilation (such as a ventilator) in the 28 days following the start of treatment.
SOFA score | day 0，day 5-7
  The SOFA score uses six criteria to reflect the function of organ systems (respiratory, blood, liver, cardiovascular, nervous, and kidney) and sets each on a score of 0-4. The objective was to describe the occurrence, development and incidence of MODS
APACHE II score | day 0，day 5-7
  The APACHE II score is based on 12 physiological indicators, age, and health status on a scale of 0-71. The higher the score, the more severe the reaction condition, the worse the prognosis, and the higher the expected fatality rate

OTHER OUTCOMES:
Blood routine test | day 0，7 day after treatment
  It mainly includes WBC, percentage of neutrophils，The percentages of white blood cells and neutrophils represent inflammation, with higher values indicating higher inflammation.
C-reactive protein | day 0，7 day after treatment
  C-reactive protein on behalf of the inflammation, the higher the value, the higher the inflammatory conditions.
Procalcitonin | day 0，7 day after treatment
  Procalcitonin, the degree of its increase is positively correlated with the degree of infection. Used in the identification of bacteria and viruses, to monitor the severity of the infection, is used to evaluate the therapeutic effect and prognosis of infection.
TNF-α | day 0，7 day after treatment
  It is one of the cytokines involved in the inflammatory response and is used to evaluate the therapeutic effect and prognosis of infection.
interleukin-6 (IL-6), interleukin-10 (IL-10) | day 0，7 day after treatment
  It is one of the cytokines involved in the inflammatory response and is used to evaluate the therapeutic effect and prognosis of infection.
Routine biochemical tests | day 0，7 day after treatment
  Among them, abnormal total bilirubin, direct bilirubin, indirect bilirubin, AST, and ALT indicated liver function problems, abnormal BNP and TnI indicated heart function problems, and abnormal creatinine and urea nitrogen indicated renal function problems
Arterial lactic acid | day 0，7 day after treatment
  Arterial lactate was significantly associated with inflammation. Inflammatory reaction period, memory increased plasma lactate levels, lactic acid leels may aggravate the inflammatory response at the same time
Thrombin time | day 0，7 day after treatment
  Its numerical and coagulation index significantly correlated, prothrombin time is screening test of the extrinsic coagulation pathway.
Partial activated thromboplastin time | day 0，7 day after treatment
  Its value is significantly correlated with coagulation indexes, and it is the most sensitive and commonly used screening test for endogenous coagulation system.
Immune function | day 0，7 day after treatment
  It mainly includes the absolute number of lymphocytes, the number of CD4+T cells, the number of CD8+T cells, the number of B cells, the number of NK cells and other indicators to evaluate the immune function of patients
Adverse event table | Day 0，7 day after treatment，14 day after treatment，28 day after treatment
  Patient safety during treatment was assessed by the Adverse Events Table
Changes in bile acid profile composition | Day 0, day 5-7
  Blood samples were collected, and the changes in the number and concentration of bile acids in the blood were analyzed to explore the changes in the composition of the bile acid spectrum before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wu JianNong, doctor, Study Chair — The First Affiliated Hospital of Zhejiang Chinese Medical University; Liu Shan, doctor, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University; Feng DanDan, master, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen MY, Li ZJ, Feng DD, Yang DD, Liu S, Fu YH, Fang BJ, Wu JN. Shenhuang Granules for patients with sepsis: study protocol of a multicenter, randomized, double-blind, placebo-controlled clinical trial. Front Med (Lausanne). 2025 Nov 21;12:1700749. doi: 10.3389/fmed.2025.1700749. eCollection 2025. PMID 41357500

DOCUMENTS (1):
  • Informed Consent Form (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT06514339/ICF_000.pdf